CLINICAL TRIAL: NCT05324059
Title: Confirmatory Study of Efficacy and Safety of the Pregabalin/Tramadol Combination Versus Pregabalin in the Management of Acute Pain of Neuropathic Origin.
Brief Title: Efficacy and Safety of Pregabalin/Tramadol Combination Versus Pregabalin in Acute Pain of Neuropathic Origin
Acronym: LOBUXALIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30901-III-21 (2)
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Neuropathic Pain
Keywords: Acute pain; Neuropathic; Pregabalin; Tramadol
MeSH Terms: conditions — Neuralgia; Acute Pain | interventions — Pregabalin; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Pregabalin/Tramadol (Experimental): Fixed dose combination tablet of 75 mg Pregabalin and 50 mg of Tramadol, orally, every 12 hours.
  Interventions: Drug: Pregabalin 75mg/ Tramadol 50 mg
- Group B: Pregabalin (Active Comparator): Monotherapy with 75 mg of Pregabalin, orally, every 12 hours.
  Interventions: Drug: Pregabalin 75mg

INTERVENTIONS:
Drug: Pregabalin 75mg/ Tramadol 50 mg — Pharmaceutical Form: Tablet Dosage: 75 mg / 50 mg Administration way: oral
  Other Names: LOBUXAL
  Arms: Group A: Pregabalin/Tramadol
Drug: Pregabalin 75mg — Pharmaceutical Form: Capsule Dosage: 75 mg Administration way: oral
  Other Names: Pregabalin
  Arms: Group B: Pregabalin

SUMMARY:
Phase IIIb confirmatory study of efficacy and safety, longitudinal, multicenter, randomized, double-blind study of the combination Pregabalin/Tramadol versus Pregabalin in the management of acute pain of neuropathic origin.

DETAILED DESCRIPTION:
Study to evaluate the efficacy and safety of the fixed-dose combination of Pregabalin/Tramadol versus Pregabalin in the management of acute pain of neuropathic origin. Patients who meet the inclusion criteria of the protocol and start treatment with the combination Pregabalin / Tramadol (75 mg / 50 mg) or Pregabalin 75 mg will be included. To evaluate the proportion of subjects who reported a success rate in the reduction of pain by 50%, the percentage of change in the pain intensity reported through the Visual Analog Pain Scale (VAS) will be calculated. This percentage will be categorized and the proportion of patients per treatment group will quantify. Changes in pain intensity during the intervention will be evaluated with the fixed-dose combination of Pregabalin/Tramadol (75 mg / 50 mg) or Pregabalin 75 mg, comparing the average difference in pain reported through VAS at days 1, 3, 5, 7, 10, 13 and 15 with respect to their baseline measurement. The mean change in reported neuropathic pain intensity across the DN4 questionnaire will also be evaluated, comparing its measurement on day 3, 10 and 15 with respect to the baseline, in each treatment group.

At visit 1 (day 3) the need for dose escalation will be evaluated (Pregabalin/Tramadol (150 mg / 50 mg) or pregabalin (150 mg)) in both treatment groups, continuing with its follow-up in the evaluation of the intensity of pain reported by EVA and DN4. The proportion of subjects who started on the dose of Pregabalin / Tramadol (75 mg / 50 mg) or Pregabalin 75 mg, those that required adjustment of dose to treatment (Pregabalin / Tramadol (150 mg / 50 mg) or Pregabalin (75 mg)), as well as the proportion of patients who suspended the treatment.

The percentage of adherence to the intervention by treatment group will be reported.

The proportion of adverse events presented during the conduct of the study will be evaluated, regardless of the dose administered, to all the subjects who have received at least one dose of the investigational drug Which will be reported be reported through frequencies and percentages and classified according to frequency, gravity, severity (intensity) and the causality of the clinical manifestation.

ELIGIBILITY:
Inclusion Criteria:

* Any gender.
* That the subject agrees to participate in the study and give its informed consent in writing.
* Age >18 years and ≤65 years of age at the start of the study.
* Neuropathic Pain Questionnaire (DN4) ≥ 4.
* Patients with proven tolerability (absence of moderate-serious adverse events) to pregabalin, defined by consumption of pregabalin 50 mg/day for 3 days.
* Women of childbearing age who have an acceptable method of contraception (eg barrier, oral hormonal, injectable, subdermal).

Exclusion Criteria:

* Contraindication and known hypersensitivity to the use of pregabalin and/or tramadol.
* The patient is participating in another clinical study involving an investigational treatment or participated in any in the previous 4 weeks.
* In the medical opinion, a disease that affects the prognosis and prevents outpatient management, for example, but not limited or restricted to: terminal cancer, heart failure, obstruction gastrointestinal including paralytic ileus, suspected surgical abdomen, respiratory failure with scheduled surgical or hospital procedures.
* Positive pregnancy test, women who are pregnant, nursing or planning a pregnancy during the conduct of the study.
* Patients with a diagnosis of respiratory diseases: status asthmaticus, asthma, chronic obstructive pulmonary disease (COPD), cor pulmonale, acute respiratory depression, hypercapnia.
* Patients who are receiving monoamine oxidase inhibitors (MAOIs) or who have received within the last 2 weeks.
* Patients with a history of seizure disorders, epileptic status, and grand mal seizures.
* Patients with a history of severe depression of the central nervous system due to consumption of opiates.
* History of acute intoxications with hypnotics, opioid analgesics and psychotropics.
* History of alcohol or drug abuse (including opiates) in the last year according to DSM-V.
* Patients with a history of severe head trauma and/or brain edema.
* History/presence of any disease or condition which, in the opinion of the Investigator, could pose a risk to the patient or confound the efficacy and safety results of the study.
* Patients with symptoms suggestive of active COVID-19 infection (i.e., fever, cough, dyspnea) and/or contact in the last 14 days with a suspected or positive patient for COVID-19.
* Patients whose participation in the study may be influenced (employment relationship with the center investigator or sponsor, inmates, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a success rate of >50% in pain reduction | 15 days
  Evaluate the proportion of subjects who reported a success rate of >50% in pain reduction at completion of the intervention, measure by the VAS (Visual Analog Scale) per treatment group. In a straight 10 centimeter line in which one end means no pain and the other end means the worst pain imaginable, the participants mark the amount of pain feeling at that moment.
Mean change in pain intensity by VAS (Visual Analog Scale) | Baseline,1,3,5,7,10, 13 and 15 days
  Evaluate the mean change in pain intensity reported on days 1, 3, 5, 7, 10, 13, and 15 with respect to its baseline measurement, reported through the VAS (Visual Analog Scale) per treatment group. In a straight 10 centimeter line in which one end means no pain and the other end means the worst pain imaginable, the participants mark the amount of pain feeling at that moment.
Mean change in pain intensity by DN4 questionnaire | Baseline, 3, 10 and 15 days
  Evaluate the mean change in pain intensity reported on days 3, 10 and 15 with respect to its baseline measurement according to the DN4 Questionnaire by treatment group.
Proportion of subjects requiring dose escalation | Day 3
  Evaluate the proportion of subjects who required dose escalation (from Pregabalin/Tramadol 75mg/50 to 150 mg/ 50 mg or Pregabalin 75mg to 150 mg, as appropriate) during the intervention, by treatment group.
Frequency of adverse events | 15 days
  Compare the frequency of adverse events presented during the study between the treatment groups.
Intensity of adverse events. | 15 days
  Compare the intensity of adverse events presented by treatment group.

SECONDARY OUTCOMES:
Adherence percentage | 15 days
  Report the percentage of adherence to the intervention by treatment group, using the count of tablets returned to the research site

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Suárez Otero, M.D, Principal Investigator — Independent consultant; Isabel E Rucker, M.D, Principal Investigator — Clinical Research Institute; Luis R Partida, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V.; Alfonso Hernández Zepeda, M.D, Principal Investigator — IMACEN S.A. de C.V.; Ma. Dolores Alonso Martínez, M.D, Principal Investigator — CICMEX, Centro de Investigación Clínica de México S. de R.L de C.V.
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor RS. Epidemiology of refractory neuropathic pain. Pain Pract. 2006 Mar;6(1):22-6. doi: 10.1111/j.1533-2500.2006.00054.x. PMID 17309705
- [Background] Torrance N, Smith BH, Bennett MI, Lee AJ. The epidemiology of chronic pain of predominantly neuropathic origin. Results from a general population survey. J Pain. 2006 Apr;7(4):281-9. doi: 10.1016/j.jpain.2005.11.008. PMID 16618472
- [Background] Matthiesen T, Wohrmann T, Coogan TP, Uragg H. The experimental toxicology of tramadol: an overview. Toxicol Lett. 1998 Mar 16;95(1):63-71. doi: 10.1016/s0378-4274(98)00023-x. PMID 9650647
- [Background] Randinitis EJ, Posvar EL, Alvey CW, Sedman AJ, Cook JA, Bockbrader HN. Pharmacokinetics of pregabalin in subjects with various degrees of renal function. J Clin Pharmacol. 2003 Mar;43(3):277-83. doi: 10.1177/0091270003251119. PMID 12638396
- [Background] Ardakani YH, Rouini MR. Pharmacokinetics of tramadol and its three main metabolites in healthy male and female volunteers. Biopharm Drug Dispos. 2007 Dec;28(9):527-34. doi: 10.1002/bdd.584. PMID 17891748
- [Background] de Moraes NV, Lauretti GR, Lanchote VL. Effects of type 1 and type 2 diabetes on the pharmacokinetics of tramadol enantiomers in patients with neuropathic pain phenotyped as cytochrome P450 2D6 extensive metabolizers. J Pharm Pharmacol. 2014 Sep;66(9):1222-30. doi: 10.1111/jphp.12255. Epub 2014 Apr 10. PMID 24717054
- [Background] Bockbrader HN, Radulovic LL, Posvar EL, Strand JC, Alvey CW, Busch JA, Randinitis EJ, Corrigan BW, Haig GM, Boyd RA, Wesche DL. Clinical pharmacokinetics of pregabalin in healthy volunteers. J Clin Pharmacol. 2010 Aug;50(8):941-50. doi: 10.1177/0091270009352087. Epub 2010 Feb 10. PMID 20147618
- [Background] Chew ML, Plotka A, Alvey CW, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pharmacokinetics of pregabalin controlled-release in healthy volunteers: effect of food in five single-dose, randomized, clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):617-26. doi: 10.1007/s40261-014-0211-4. PMID 25078976
- [Background] Lee S, Kim Y, Lee JJS, Im G, Cho JY, Chung JY, Yoon S. A pharmacokinetic drug-drug interaction study between pregabalin and tramadol in healthy volunteers. Eur J Clin Pharmacol. 2018 Dec;74(12):1605-1613. doi: 10.1007/s00228-018-2543-0. Epub 2018 Aug 22. PMID 30136102
- [Background] Vandenbossche J, Richards H, Solanki B, Van Peer A. Single- and multiple-dose pharmacokinetic studies of tramadol immediate-release tablets in children and adolescents. Clin Pharmacol Drug Dev. 2015 May-Jun;4(3):184-92. doi: 10.1002/cpdd.169. Epub 2014 Dec 22. PMID 27140798
- [Background] Vandenbossche J, Van Peer A, Richards H. Single-Dose Pharmacokinetic Study of Tramadol Extended-Release Tablets in Children and Adolescents. Clin Pharmacol Drug Dev. 2016 Sep;5(5):343-53. doi: 10.1002/cpdd.266. Epub 2016 Jun 12. PMID 27138295
- [Background] Dou Z, Jiang Z, Zhong J. Efficacy and safety of pregabalin in patients with neuropathic cancer pain undergoing morphine therapy. Asia Pac J Clin Oncol. 2017 Apr;13(2):e57-e64. doi: 10.1111/ajco.12311. Epub 2014 Dec 22. PMID 25530068
- [Background] Harati Y, Gooch C, Swenson M, Edelman S, Greene D, Raskin P, Donofrio P, Cornblath D, Sachdeo R, Siu CO, Kamin M. Double-blind randomized trial of tramadol for the treatment of the pain of diabetic neuropathy. Neurology. 1998 Jun;50(6):1842-6. doi: 10.1212/wnl.50.6.1842. PMID 9633738
- [Background] Wang SL, Wang H, Nie HY, Bu G, Shen XD, Wang H. The efficacy of pregabalin for acute pain control in herpetic neuralgia patients: A meta-analysis. Medicine (Baltimore). 2017 Dec;96(51):e9167. doi: 10.1097/MD.0000000000009167. PMID 29390451
- [Background] Markman J, Resnick M, Greenberg S, Katz N, Yang R, Scavone J, Whalen E, Gregorian G, Parsons B, Knapp L. Efficacy of pregabalin in post-traumatic peripheral neuropathic pain: a randomized, double-blind, placebo-controlled phase 3 trial. J Neurol. 2018 Dec;265(12):2815-2824. doi: 10.1007/s00415-018-9063-9. Epub 2018 Sep 21. PMID 30242745
- [Background] Onakpoya IJ, Thomas ET, Lee JJ, Goldacre B, Heneghan CJ. Benefits and harms of pregabalin in the management of neuropathic pain: a rapid review and meta-analysis of randomised clinical trials. BMJ Open. 2019 Jan 21;9(1):e023600. doi: 10.1136/bmjopen-2018-023600. PMID 30670513
- [Background] Freynhagen R, Serpell M, Emir B, Whalen E, Parsons B, Clair A, Latymer M. A comprehensive drug safety evaluation of pregabalin in peripheral neuropathic pain. Pain Pract. 2015 Jan;15(1):47-57. doi: 10.1111/papr.12146. Epub 2013 Nov 27. PMID 24279736
- [Background] Mercier F, Claret L, Prins K, Bruno R. A Model-Based Meta-analysis to Compare Efficacy and Tolerability of Tramadol and Tapentadol for the Treatment of Chronic Non-Malignant Pain. Pain Ther. 2014 Jun;3(1):31-44. doi: 10.1007/s40122-014-0023-5. Epub 2014 Feb 13. PMID 25135386
- [Background] Blanco E, Galvez R, Zamorano E, Lopez V, Perez M. [Prevalence of neuropathic pain according to the NP4 test in primary care]. Semergen. 2012 May-Jun;38(4):203-10. doi: 10.1016/j.semerg.2011.10.012. Epub 2011 Dec 21. Spanish. PMID 23544720
- [Background] Moon DE, Lee DI, Lee SC, Song SO, Yoon DM, Yoon MH, Kim HK, Lee YW, Kim C, Lee PB. Efficacy and tolerability of pregabalin using a flexible, optimized dose schedule in Korean patients with peripheral neuropathic pain: a 10-week, randomized, double-blind, placebo-controlled, multicenter study. Clin Ther. 2010 Dec;32(14):2370-85. doi: 10.1016/j.clinthera.2011.01.014. PMID 21353106
- See also: Rincon Carvajal AM, Olaya Osorio CA, Martínez Rojas S, Ibata Bernal L. Recommendations based on in evidence for the management of neuropathic pain in Primary Health Care (Review of the literature). Rev Soc Esp Pain [Internet]. 2018 [cited 2021 Dec 29]; — http://gestoreditorial.resed.es/DOI/PDF/ArticuloDOI_3673.pdf
- See also: Health Secretary. Official Mexican STANDARD NOM-220-SSA1-2016, Installation and operation of the pharmacovigilance — http://dof.gob.mx/nota_detalle.php?codigo=5490830&fecha=19/07/2017.